## **Cover Page**

## **Statistical Analysis Plan**

Study Title: Unilateral Strength Training and Mirror Therapy for Patients with Chronic

**Stroke: A Pilot Randomised Controlled** 

Trial Document creation date: July 12th 2015

NCT number [not yet assigned].

Identifiers: [NCT ID not yet assigned]

Statistical Analysis Plan for Unilateral Strength Training and Mirror Therapy for Patients with Chronic Stroke: A Pilot Randomised Controlled Trial (Daniel Simpson, IT Sligo)

Data was analysed using IBM SPSS for Windows (Version 20, Chicago, IL, USA). All variables were tested for normal distribution using the Shapiro-Wilk test. Sample demographics and outcome measures are described in Mean±SD. Between group differences for demographic characteristics were tested for using the Independent t test, the Mann-Whiteny U test and the Chi Square test. Within group means (T1 v T2 and T1 v T3) were analysed using the Paired-Samples-t-test for normally distributed data and the Wilcoxon Signed Rank test for non-normally distributed data. Between group differences (ST v MST) in change over the intervention were tested for using the independent-sample-t-test (normal distribution) and the Mann-Whitney U test (non-normal distribution or non-continuous scale). A *p*-value <0.05 was considered statistically significant and effect sizes expressed as either Cohen's d or *r*. Effect size for within group differences were calculated as follows:

Paired differences effect size =  $\frac{mean}{Sd}$  or  $r=Z/\sqrt{n}$ . Effect sizes for between group differences for the independent-samples-t-test were calculated using and expressed as Cohen's d. For the Mann-Whitney U test, between group differences were calculated as  $r=Z/\sqrt{n}$ .